CLINICAL TRIAL: NCT02119442
Title: Transcatheter Valve Implantation in Patients With Dysfunctional Left and Right Sided Heart Valves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jamil Aboulhosn, Associate Professor of Clinical Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-001008
Record Dates: First submitted 2014-04-08; First posted 2014-04-21 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Eisenmenger Syndrome
Keywords: Eisenmenger Syndrome, Pulmonary Arterial Hyptertension
MeSH Terms: conditions — Eisenmenger Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcatheter Valve Implantation (Other): Intervention, Transcatheter Valve Implantation with Melody or Sapien bioprosthetic valve Standard of care intervention.
  Interventions: Device: Transcather Valve Implantation

INTERVENTIONS:
Device: Transcather Valve Implantation — Transcather Valve Implantation
  Other Names: Medtronic Melody Transcatheter Valve; Melody TPV 20 PB1016:Melody TPV 22 PB1018; Edwards SAPIEN Transcatheter Heart Valve

SUMMARY:
A growing body of data, suggests that transcatheter valves are effective when implanted in other locations (mitral, aortic, tricuspid) and in high pressure environments. The investigators plan to offer transcatheter valve implantation as an alternative to high risk surgery in patients who require revision of a stenotic or regurgitant valve in the non-pulmonary position (mitral, aortic, tricuspid). This therapy can provide an alternative to patients who may be considered high risk and may not be able to survive a surgical procedure.The use of the devices on this protocol are for medical treatment and are not part of a clinical trial.

DETAILED DESCRIPTION:
Many forms of congenital and structural heart disease require surgical placement of prosthetic valves and conduits. These conditions include many common congenital heart abnormalities such as Tetralogy of Fallot, Double Outlet Right Ventricle, Truncus Arteriosus and patients who require the Ross procedure for aortic stenosis. There are a variety of acquired conditions, including calcific aortic valve stenosis that may require surgical or transcatheter valve treatment. Unfortunately, when valved conduits are placed surgically, they ultimately become narrowed or regurgitant and require periodic replacement. Thus, patients with these conditions often undergo multiple open heart surgeries during their lifetime. Although the risk of mortality with this kind of surgery is low, surgical intervention is associated with significantly longer recovery times and more patient discomfort when compared to transcatheter interventions. Over the last decade, techniques have been developed to palliate these forms of congenital and structural heart disease using catheters inserted through blood vessels in the groin. These transcatheter techniques have allowed patients to delay or avoid open heart surgery.

The Medtronic Melody Trancatheter Valve and the Edwards SAPIEN Transcatheter Heart Valve are both bioprosthetic valves mounted within metal stents. Their entire structure is collapsible, allowing it to be inserted through delivery sheaths and threaded into the heart, typically without the need of surgical cardiopulmonary bypass. Some of these procedures may be performed using a hybrid technique of minimal surgical access and transcatheter valve delivery. The valves can then be expanded into place by inflating a balloon (similar to how stents are placed elsewhere in the heart, like the coronary artery). The Melody Valve received a humanitarian device exemption (HDE) from the FDA and the Edwards Sapien Valve has market approval from the FDA.The investigators plan to offer these transcatheter valves as alternatives to eligible patients who require replacement of a stenotic or regurgitant valve in all left and right sided positions.

The intended role of the Melody Transcatheter Pulmonary Valve is to restore pulmonary valve function in patients with a dysfunctional RVOT conduit and a clinical indication for pulmonary valve replacement. Unlike currently available options for pulmonary valve replacement, the TPV is intended to be placed with a transcatheter delivery system, and thus does not require surgical incisions, open heart surgery, cardiopulmonary bypass, or the various morbidities associated with surgical pulmonary valve replacement. The Edwards Sapien Valve is delivered in the same manner, but was intended for use in the aortic position. The ultimate goals and durability of the TPV may differ among patients with different indications. At a minimum, the intention is that the TPV will improve hemodynamic function, mitigate the adverse impact of valve regurgitation and/or obstruction, and effectively extend the longevity of the existing conduit and defer or obviate the need for conduit replacement. These techniques may decrease the number of open heart surgeries required over the course of a patient's lifetime, thereby decreasing the cumulative morbidity and risk associated with such operations.

With regards to valve replacement in any position with an adequate landing zone, the Melody Valve and Edwards Sapien Valve are presently being utilized at multiple United States centers for valve replacement in all positions in patients who are considered high risk candidates for surgical valve replacement. A recent article published by Zahn et al reported an experience in tricuspid valve implantations at three United States centers and one Austrailian center. Procedural success was achieved in all patients. Tricuspid regurgitation was reduced to mild or none in all patients. Noted complications were consistent with known risks of cardiac catheterization and Melody Valve implantation, regardless of indication. Similarly, an article published by Kenny et al demonstrated the successful implantation of the Sapien valve in the tricuspid position. Gillespie et al, recently published a series of Melody implants in the mitral position in sheep that had undergone annuloplasty ring placement. Other investigators have successfully implanted the Melody valve in the aortic and mitral positions in patients with good immediate and short/intermediate term outcomes (Ben-Gal et al, Hasan et al, Gossl et al). The Edwards Sapien Valve has several reports of positive outcomes when implanted within the aortic position (Thomas et al, Moat et al, Webb et al) and two case series that report encouraging results when placed in the mitral position. (Seiffert et al, Cheung et al)

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered eligible for transcatheter valve implantation if the risk of serious morbidity or mortality with surgical intervention is deemed to be greater than 10 percent by the treating cardiologist and consulting surgeon. The Melody Valve is intended for use in the following clinical conditions:
* Existence of a full (circumferential) RVOT conduit that was equal to or greater than 16 mm in diameter when originally implanted, AND
* Dysfunctional RVOT conduits with a clinical indication for intervention, AND EITHER
* Regurgitation ≥ moderate
* Stenosis: mean right ventricular outflow tract gradient ≥ 35 mmHg
* The Edwards Sapien Valve will be used in the aortic position for valves and conduits larger than 23mm in diameter with a landing zone less than 26-27mm, otherwise the melody valve will be considered
* The Edwards Sapien Vavle will also be considered in other positions that have an adequate landing zone and a large enough circumference
* The Melody valve may be utilized outside of its approved indications for valve replacement in high risk surgical patients

Exclusion Criteria:

* There are no known contraindications for implantation of the Melody Valve or the Edwards Sapien Valve

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil A Aboulhosn, MD, FACC, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Kondo N, Shuto T, McGarvey JR, Koomalsingh KJ, Takebe M, Gorman RC, Gorman JH 3rd, Gillespie MJ. Melody valve-in-ring procedure for mitral valve replacement: feasibility in four annuloplasty types. Ann Thorac Surg. 2012 Mar;93(3):783-8. doi: 10.1016/j.athoracsur.2011.12.021. PMID 22364973
- [Background] Riede FT, Dahnert I. Implantation of a Melody valve in tricuspid position. Catheter Cardiovasc Interv. 2012 Sep 1;80(3):474-6. doi: 10.1002/ccd.23404. Epub 2012 Mar 14. PMID 22105855
- [Background] Ben-Gal Y, Finkelstein A, Bruckheimer E, Banai S, Keren G, Kramer A, Uretzky G. Transapical implantation of a Melody valve in a degenerated low-diameter prosthetic aortic valve. Circulation. 2013 Apr 23;127(16):e553-6. doi: 10.1161/CIRCULATIONAHA.112.127027. No abstract available. PMID 23609553
- [Background] Cheung AW, Gurvitch R, Ye J, Wood D, Lichtenstein SV, Thompson C, Webb JG. Transcatheter transapical mitral valve-in-valve implantations for a failed bioprosthesis: a case series. J Thorac Cardiovasc Surg. 2011 Mar;141(3):711-5. doi: 10.1016/j.jtcvs.2010.11.026. Epub 2011 Jan 26. PMID 21269643
- [Background] Kenny D, Hijazi ZM, Walsh KP. Transcatheter tricuspid valve replacement with the Edwards SAPIEN valve. Catheter Cardiovasc Interv. 2011 Aug 1;78(2):267-70. doi: 10.1002/ccd.23016. Epub 2011 Jul 15. PMID 21766424

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcatheter Valve Implantation: Intervention, Transcatheter Valve Implantation with Melody or Sapien bioprosthetic valve Standard of care intervention. All participants were considered to be under the same Arm/Group.
  Transcather Valve Implantation: Transcather Valve Implantation
Period: Overall Study
Arm/Group | Transcatheter Valve Implantation
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcatheter Valve Implantation
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 62
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 25 [3 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Infective Endocarditis
Description: The investigator will be assessing the efficacy of transcatheter heart valve (THV) by evaluating survival and development of infective endocarditis as an adverse event.
Time Frame: 8 years
Measure: Number; unit: participants
Arm/Group | Transcatheter Valve Implantation
Number analyzed (Participants) | 90
participants | 9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until the latest follow up time point that the patients were seen by a physician. This time point included at least one year of follow up or more.
Arm/Group | Transcatheter Valve Implantation
All-Cause Mortality (participants affected / at risk) | 4/90
Serious Adverse Events (participants affected / at risk) | 9/90
Other Adverse Events (participants affected / at risk) | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcatheter Valve Implantation (N=90)
infective endocarditis (Cardiac disorders) | 9 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-10-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT02119442/SAP_000.pdf
  • Study Protocol (2013-08-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT02119442/Prot_001.pdf